CLINICAL TRIAL: NCT04883788
Title: The Impact of COVID-19 Pandemic on the Nursing-sensitive and Rehabilitation Outcomes of Patients Undergoing Hip or Knee Replacement: a Single Centre Retrospective Study
Brief Title: The Impact of COVID-19 Pandemic on Hip and Knee Replacement
Acronym: PTA/PTGCovid
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Mattia Morri, Physiotherapist, Istituto Ortopedico Rizzoli
Other Study IDs: Codice AVEC 352/2021/Oss/IOR
Record Dates: First submitted 2021-05-11; First posted 2021-05-12 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Covid19; Hip Arthropathy; Knee Arthropathy
Keywords: Covid19 pandemic; Hip Arthropathy; Knee Arthropathy; Nursing Sensitive Outcome; Rehabilitation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pandemic group: Patients undergone hip and knee replacement during pandemic period (June-december 2020)
  Interventions: Other: Pandemic period
- Pre-pandemic group: Patients undergone hip and knee replacement during the pre-pandemic period (january-march 2020)

INTERVENTIONS:
Other: Pandemic period — Perioperative care (nursing and physiotherapy) provided to patients treated with hip and knee replacement during the pandemic period
  Groups: Pandemic group

SUMMARY:
During the COVID-19 pandemic, the care of patients undergoing hip or knee replacement for osteoarthritis remains a clinical priority. To date, there is limited empirical knowledge about the impact of pandemic on the care of patients surgically treated for orthopaedic diseases, affected or not by COVID-19.

The aim of the present study is to describe and investigate the effects of the COVID-19 pandemic on the nursing-sensitive and rehabilitation outcomes of patients undergoing hip and knee replacement.

DETAILED DESCRIPTION:
From hospital electronic registry of patients will be possible to screen the patients eligible for the study.

From each electronic patients record, health professional researchers will be responsable to collect data.

Variables about nursing and physiotherapy care, the staffing activities and the outcome achieved by the patients will be collected.

To investigate the impact of COVID-19 pandemic, data of the pandemic period (june-december 2020), will be compared with the data of the same year pre-pandemic (january-march 2020). During the period from april to may 2020, only orthopaedic surgery for emergency trauma or disease was allowed.

ELIGIBILITY:
Inclusion Criteria:

Patients undergone hip or knee replacement for osteoarthritis

Exclusion Criteria:

Patients undergone hip or knee replacement for fracture, trauma or oncological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undegone hip or knee replacement for osteoarthrits during 2020
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
early independence | 5 days after surgery
  The recovery of patients of the independence measured by ILOA score
early ambulation | during hospitalization
  The first time that the patient is able to walk with elbow crutches after surgery

SECONDARY OUTCOMES:
early upstairs | during hospitalization
  The first time that the patient is able to upstairs after surgery
Wound infection | during hospitalization
  Incidence of wound infection
Urinary infections | during hospitalization
  Incidence of urinary infection
Pressure ulcers | during hospitalization
  Incidence of pressure ulcers
Paralytic ileus | during hospitalization
  diagnosis or sign of paralytic ileus

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aiken LH, Sloane D, Griffiths P, Rafferty AM, Bruyneel L, McHugh M, Maier CB, Moreno-Casbas T, Ball JE, Ausserhofer D, Sermeus W; RN4CAST Consortium. Nursing skill mix in European hospitals: cross-sectional study of the association with mortality, patient ratings, and quality of care. BMJ Qual Saf. 2017 Jul;26(7):559-568. doi: 10.1136/bmjqs-2016-005567. Epub 2016 Nov 15. PMID 28626086
- [Background] Randau TM, Jaenisch M, Haffer H, Schomig F, Kasapovic A, Olejniczak K, Flechtenmacher J, Perka C, Wirtz DC, Pumberger M. Collateral effect of COVID-19 on orthopedic and trauma surgery. PLoS One. 2020 Sep 8;15(9):e0238759. doi: 10.1371/journal.pone.0238759. eCollection 2020. PMID 32898179
- [Background] Wong JSH, Cheung KMC. Impact of COVID-19 on Orthopaedic and Trauma Service: An Epidemiological Study. J Bone Joint Surg Am. 2020 Jul 15;102(14):e80. doi: 10.2106/JBJS.20.00775. PMID 32675668
- [Background] Macey ARM, Butler J, Martin SC, Tan TY, Leach WJ, Jamal B. 30-day outcomes in hip fracture patients during the COVID-19 pandemic compared to the preceding year. Bone Jt Open. 2020 Nov 2;1(7):415-419. doi: 10.1302/2633-1462.17.BJO-2020-0077.R1. eCollection 2020 Jul. PMID 33215132
- [Background] Shields RK, Enloe LJ, Evans RE, Smith KB, Steckel SD. Reliability, validity, and responsiveness of functional tests in patients with total joint replacement. Phys Ther. 1995 Mar;75(3):169-76; discussion 176-9. doi: 10.1093/ptj/75.3.169. PMID 7870749